CLINICAL TRIAL: NCT00253149
Title: The Safety And Efficacy Of Risperdal� (Risperidone) Versus Placebo Versus Haloperidol As Add-On Therapy To Mood Stabilizers In The Treatment Of The Manic Phase Of Bipolar Disorder
Brief Title: A Study of the Effectiveness and Safety of Risperidone as add-on Therapy to Mood Stabilizers in the Treatment of Manic Episodes Associated With Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006040
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Bipolar Disorders; Manic Disorder
Keywords: risperidone; antipsychotic agents; bipolar disorders; manic episode
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of risperidone (an antipsychotic medication) versus placebo as add-on therapy to mood stabilizers in the treatment of manic episodes associated with bipolar disorder.

DETAILED DESCRIPTION:
Risperidone, widely used in the treatment of schizophrenia, has been shown to be effective in the treatment of manic and mixed episodes associated with bipolar disorders. Antipsychotic drugs like risperidone have also been used as additional therapeutic agents in the treatment of patients who are not responsive to mood stabilizers alone. This is a randomized, double-blind, placebo-controlled study to evaluate the effectiveness and safety of risperidone compared with placebo, as an addition to mood stabilizing drugs in the treatment of patients experiencing manic episodes. Treatment of one group of patients with haloperidol is used as an internal control in the trial. The study has two phases: a double-blind treatment phase (3 weeks) and an open-label phase (10 weeks). During the double-blind treatment phase patients receive risperidone, haloperidol, or placebo tablets to be taken once a day at gradually increasing doses (adjusted to 1 to 6 mg/day for risperidone and 2 to 12 mg/day for haloperidol), while continuing treatment with a mood stabilizer (lithium or valproate). In the open-label phase all patients receive risperidone with the dosage gradually adjusted to achieve optimal effectiveness (dose range of 0 to 6 mg/day); in this phase patients continue therapy with a mood stabilizer (lithium, valproate, or, for this phase only, carbamazepine). The primary measure of effectiveness is the change in the Young Mania Rating Scale (YMRS) total score from baseline to end of double-blind treatment. Additional assessments of effectiveness include the Brief Psychiatric Rating Scale (BPRS); the Clinical Global Impression (CGI), which evaluates the change in severity of the disorder; and the Hamilton Depression Rating Scale (HAMD). Safety assessments include the incidence of adverse events throughout the study; measurement of vital signs (pulse and blood pressure) and evaluation of the presence and severity of extrapyramidal symptoms by the Extrapyramidal Symptom Rating Scale (ESRS) at specified intervals; and clinical laboratory tests (hematology, biochemistry, urinalysis) before study initiation, at completion of double-blind treatment, and at the end of study. The study hypothesis is that daily treatment with risperidone as add-on therapy provides better effectiveness than placebo, as measured by Young Mania Rating Scale scores, in the treatment of the manic phase of bipolar disorder. Double-blind (daily doses, taken orally once a day) - Days 1 and 2: risperidone 2 mg, haloperidol 4 mg, or placebo. Days 3 and 4: risperidone 1 - 4 mg, haloperidol 2 - 8 mg, or placebo. Days 5 - 21: risperidone 1 - 6 mg, haloperidol 2 - 21 mg, or placebo. Open-label: risperidone 0 - 6 mg/day for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar Disorder according to Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV)
* hospitalized for mania with a score >=20 on the Young Mania Rating Scale (YMRS) (patients with concurrent symptoms of depression are eligible)
* inpatient for a minimum of the first 4 days of double-blind treatment
* therapy with lithium or valproate (mood stabilizers) at start of treatment with study medication
* medically stable on the basis of physical examination, medical history, and electrocardiogram results.

Exclusion Criteria:

* Other Axis I DSM-IV diagnosis (except nicotine or caffeine dependence)
* history of alcohol or drug abuse or dependence within 4 weeks of starting the study
* seizure disorder requiring medication
* known sensitivity to risperidone, haloperidol, lithium, valproate or carbamazepine
* pregnant or nursing females, or those lacking adequate contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Study Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
Change in Young Mania Rating Scale (YMRS) total score from baseline to end of double-blind treatment

SECONDARY OUTCOMES:
Changes from baseline to end of double-blind treatment in Brief Psychiatric Rating Scale (BPRS), Clinical Global Impression (CGI) severity, and Hamilton Depression Rating Scale (HAMD); incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Sachs GS, Grossman F, Ghaemi SN, Okamoto A, Bowden CL. Combination of a mood stabilizer with risperidone or haloperidol for treatment of acute mania: a double-blind, placebo-controlled comparison of efficacy and safety. Am J Psychiatry. 2002 Jul;159(7):1146-54. doi: 10.1176/appi.ajp.159.7.1146. PMID 12091192